CLINICAL TRIAL: NCT01592448
Title: Consumer Understanding and Use of Non-Prescription Analgesics, Investigation of Efficacy of Improved Acetaminophen Labeling
Brief Title: Investigation of Efficacy of Improved Acetaminophen Labeling
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Emory University (Other); McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Principal Investigator, Michael S. Wolf, Associate Professor, Northwestern University
Other Study IDs: McNeil-7247
Record Dates: First submitted 2011-11-28; First posted 2012-05-07 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Acetaminophen Overdose; Pain
Keywords: Acetaminophen; Patient Safety; Health Literacy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Usual Care: Participants will be shown "standard" (defined as currently commercially available) over-the-counter and prescription medicine bottles and asked questions regarding safety and use. Participants will also be shown additional "standard" over-the-counter bottles and asked whether these comparison bottles could safely be taken in addition to the primary products shown.
- Written Orientation: Participants will be exposed to over-the-counter and prescription bottles "enhanced" with an icon pertaining to active ingredient and asked questions regarding safety and use. Participants will be exposed to a flier describing the safe use of acetaminophen and orienting the participant towards the icon that is used to indicate the presence of acetaminophen in a product. This flier will be passively hanging within sight of the participant in the room, but no verbal explanation of the flier will be given to the participant. (This is designed to represent a passive education campaign such as posters in drug stores that may be used should these icons be adopted by manufacturers.)
  Interventions: Behavioral: Active Ingredient Icon
- Written + Verbal Orientation: Participants will be exposed to over-the-counter and prescription bottles "enhanced" with an icon pertaining to active ingredient and asked questions regarding safety and use. Participants will be exposed to a flier describing the safe use of acetaminophen and orienting the participant towards the icon that is used to indicate the presence of acetaminophen in a product. Research personnel will also verbally go through the flier with the participant and answer any questions in a standardized fashion. (This is designed to represent an active education campaign such as pharmacist counseling that may be used should these icons be adopted by manufacturers.)
  Interventions: Behavioral: Active Ingredient Icon

INTERVENTIONS:
Behavioral: Active Ingredient Icon — Enhanced bottles will have a symbol, or icon, designed to draw attention to active ingredient information. The icon is a black hexagon containing two letters denoting the active ingredient of the medication (i.e. "Ac" for acetaminophen). Over-the-counter bottles will have the icon placed on the front of the bottle next to active ingredient information and on the back of the bottle in the drug facts to the left of the active ingredient information. Prescription bottles will have the icon placed below the directions for how to take the medication and will be accompanied by a brief statement indicating the medicine contains acetaminophen.
  Groups: Written + Verbal Orientation; Written Orientation

SUMMARY:
The purpose of this study is to evaluate, through brief, one-on-one cognitive interviews, the efficacy of 'enhanced' acetaminophen messages and icons in improving consumer understanding and use of prescription (Rx) and non-prescription (over-the-counter, OTC) acetaminophen containing products compared to the current standard.

DETAILED DESCRIPTION:
Acetaminophen is a pain reliever and fever reducer found in many over-the-counter (OTC) analgesics as well as prescription (Rx) products commonly prescribed at discharge from the emergency department. 1 An estimated 36% of Americans ingest acetaminophen at least once a month.1, 2 While acetaminophen is generally safe and effective when used at recommended doses, acetaminophen overdose has surpassed viral hepatitis as the leading cause of acute liver failure (ALF) in the United States.2-4 Moreover, one half to two-thirds of overdoses leading to acute liver failure are unintentional, suggesting the root cause may be poor understanding of medication labeling or failure to recognize the consequences of exceeding the recommended maximum daily dosage.2-4 On-going studies by this research group have shown patient misunderstanding of dosing instructions and warnings associated with OTC medicines to be prevalent.

It has also been suggested that patients receiving prescription medications containing acetaminophen may not be informed or aware of the potential risk of acetaminophen overuse when taking prescription products in combination with over-the-counter pain relievers.1 This is supported by the finding that a third of narcotic users were simultaneously using an OTC acetaminophen containing product in a multicenter study of ALF cases.2 To address the growing concern of acetaminophen misuse, in June 2009 the US Food and Drug Administration (FDA) convened a panel to discuss the maximum dose recommendations of acetaminophen found in OTC medications. The panel concluded that there was a notable lack of available evidence on consumer understanding and use of over-the-counter acetaminophen products. Studies are needed to explore patients' 1) knowledge of potential acetaminophen overdose when using prescription analgesics simultaneously with non-prescription acetaminophen and 2) avenues available to increase awareness of potential acetaminophen overdose from misuse of both OTC and Rx acetaminophen containing medicines.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* English speaking

Exclusion Criteria:

* Visual or hearing impairments
* Moderate to severe cognitive impairments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two types of practices - an academic general medicine clinic and the other a community health center - will serve as performance sites.
Sampling Method: Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Functional Understanding and Use | 40 minutes
  Functional understanding (via teachback and demonstration) of acetaminophen label information (OTC & Rx), including 1) active ingredient, 2) maximum daily dose, and 3) risks associated with misuse.

SECONDARY OUTCOMES:
Health literacy (NVS) | 40 minutes
  The NVS (Newest Vitals Sign) is designed to provide a valid and quick assessment of participant health literacy. The assessment is based on a nutrition label from an ice cream container. Patients are given the label and then asked 6 questions about it.
Participant characteristics | 40 minutes
  Basic demographic characteristics (age, sex, race/ ethnicity), socioeconomic information (education, household income), health status information (self-reported overall health), recent medication use and beliefs about over-the-counter medicines will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Wolf, PhD, MPH, Principal Investigator — Northwestern University; Ruth M. Parker, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Grady Memorial Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Chicago LakeShore Medical Association, Chicago, Illinois
  - Mercy Hospital, Chicago, Illinois

REFERENCES:
- [Background] Fosnocht D, Taylor JR, Caravati EM. Emergency department patient knowledge concerning acetaminophen (paracetamol) in over-the-counter and prescription analgesics. Emerg Med J. 2008 Apr;25(4):213-6. doi: 10.1136/emj.2007.053850. PMID 18356351
- [Background] Larson AM, Polson J, Fontana RJ, Davern TJ, Lalani E, Hynan LS, Reisch JS, Schiodt FV, Ostapowicz G, Shakil AO, Lee WM; Acute Liver Failure Study Group. Acetaminophen-induced acute liver failure: results of a United States multicenter, prospective study. Hepatology. 2005 Dec;42(6):1364-72. doi: 10.1002/hep.20948. PMID 16317692
- [Background] Bower WA, Johns M, Margolis HS, Williams IT, Bell BP. Population-based surveillance for acute liver failure. Am J Gastroenterol. 2007 Nov;102(11):2459-63. doi: 10.1111/j.1572-0241.2007.01388.x. Epub 2007 Jun 29. PMID 17608778
- [Background] Ostapowicz G, Fontana RJ, Schiodt FV, Larson A, Davern TJ, Han SH, McCashland TM, Shakil AO, Hay JE, Hynan L, Crippin JS, Blei AT, Samuel G, Reisch J, Lee WM; U.S. Acute Liver Failure Study Group. Results of a prospective study of acute liver failure at 17 tertiary care centers in the United States. Ann Intern Med. 2002 Dec 17;137(12):947-54. doi: 10.7326/0003-4819-137-12-200212170-00007. PMID 12484709